CLINICAL TRIAL: NCT06923150
Title: A Randomised Clinical Investigation to Assess Efficacy of Low Volume Transanal Irrigation by Qufora® IrriSedo MiniGo Versus Conservative Treatment for Low Anterior Resection Syndrome Patients
Acronym: MINIGO
Status: Recruiting | Type: Observational
Sponsor: Qufora A/S (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02656-39
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gastroenterology; LARS - Low Anterior Resection Syndrome; Rectal Cancer
Keywords: LARS; Transanal Irrigation; Minigo; rectal cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TAI + SOC: Low volume TAI MiniGo + Standard of Care (SOC) conservative treatments
- SOC: Standard of Care (SOC) conservative treatments:
  dietary management, counselling, medication: anti-diarrheic or constipation treatment according to the prescription following usual practice, and food supplement excluding: suppository, ano-rectal stimulation, physiotherapy small enemas, etc…

SUMMARY:
The purpose of this post-market clinical follow up study is to assess the efficacy on clinical symptoms of LARS of low volume Transanal Irrigation by MiniGo in conjunction with conservative treatment versus conservative treatment at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged from 18 years
2. Patients electively treated for rectal cancer with a low anterior resection
3. Between 3 and 18 months after the conservative colorectal surgery or 3 and 18 months after the stoma reversal if applicable
4. LARS score >= 25 (minor or major LARS) (Emmertsen and Laurberg 2012) AND LARS definition as consensus with at least one symptom that results in at least one consequence (Keane et al. 2020)
5. Adult for whom previous conservative treatments were started for at least a month
6. Mental and physical capability of the patient to handle the MiniGo by himself.
7. Check of the anastomosis (no signs of leakage or clinical relevant stenosis) and absence of local recurrence by Rectal digital examination of the anastomosis, any other exam used in the current practice
8. Patient affiliated to the health social security system

Exclusion Criteria:

1. Contra-indication to use TAI
2. Former use of TAI (post colo-rectal surgery)
3. Clinically relevant stenosis
4. Current metastatic disease or local recurrence
5. Ongoing chemotherapy
6. Postoperative radiotherapy for rectal cancer
7. History of diarrhoeal disease
8. Inflammatory bowel disease
9. Dementia
10. Spinal cord injury, multiple sclerosis, Parkinson's disease or other significant disease assessed to be a contributory cause to LARS symptoms.
11. Patient with cancer recurrence
12. Patient with a life expectancy < 1 year
13. Participating to another clinical trial for the treatment of LARS symptom
14. Ongoing pelvic floor rehabilitation/biofeedback
15. Pregnancy or intention to become pregnant during the trial period
16. Inability and unwillingness to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: minor and major LARS patients LARS score >= 25
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
LARS score difference | 3-month follow-up
  The primary endpoint is defined by the LARS score difference between inclusion and 3-month follow-up for each randomisation group.

SECONDARY OUTCOMES:
efficacy on clinical symptom of transanal Irrigation by MiniGo in improving the LARS score at 6 weeks | 6-week follow-up
  LARS difference score between inclusion and 6-week follow-up will be calculated for each randomised arm using descriptive statistics and confidence intervals
QoL with the EORTC QLQ-C30 EORTC QLQ-CR29 | 3-month follow- up
  EORTC-QLQ-C30 and EORTC-QLQ-CR29 differences scores between inclusion and 3-month follow-up will be calculated for each randomised arm using descriptive statistics and confidence intervals.
  Also, statistical tests of superiority will be performed comparing EORTC-QLQ-C30 and EORTC-QLQ-CR29 differences between inclusion and 3-month follow-up between interventional arm and control arm
change (reduction) of symptoms and consequences | 6 weeks and 12 weeks
  To assess the number of patients showing a change (reduction) of symptoms and consequences, as stated in the consensus definition at 6 and 12 weeks The number and the proportion of patients with each item of the LARS international consensus definition at 6 and 12 weeks will be calculated.
  Also, the proportion of patients who are considered as having no LARS at 6 and 12 weeks will be calculated with a confidence interval
patient satisfaction | 6 weeks and 12 weeks
  to assess the patient satisfaction at 6 and 12 weeks, The proportion of patients satisfied by the treatment evaluated with the 5-point Likert Scale at 6 and 12 weeks will be calculated with a confidence interval.
compliance of the patient to the treatmen | 6 weeks and 12 weeks
  to assess the compliance of the patient to the treatment at 6 and 12 weeks Compliance with the treatment during the 6 and 12 weeks of study with the number of days of MiniGo use per week will be calculated using descriptive statistics and confidence intervals
incontinence anal score | 12 weeks
  To access the incontinence anal score at 12 weeks Wexner difference score between inclusion and 12-week follow-up will be calculated for each randomised arm using descriptive statistics and confidence intervals.
  Also, statistical tests of superiority will be performed comparing Wexner differences between inclusion and 12-week follow-up between interventional arm and control arm.
reduction of defecations per day and night | 6 weeks and 12 weeks
  To assess the reduction of defecations per day and night The mean number of defecations per day and per night during the week before the randomisation and the week before the follow-up visit at 6 and 12 weeks will be calculated.
time spent on bowel management (in the toilets room) | 12 weeks
  To assess the time spent on bowel management (in the toilets room) Mean times spent in the toilets room per day the week before the randomisation and the week before the follow-up visit at 12 weeks will be calculated using descriptive statistics.
patient health organization and resources needed | 12 weeks
  To evaluate the patient health organization and resources needed at 12 weeks Data about quantity of organization and resources needed (professional activities, treatment, medical and specialize consultation, home helpers) will be presented using descriptive statistics.
improving the LARS score | 6, 9 and 12 months
  to assess the efficacy on clinical symptom of Transanal Irrigation by MiniGo in improving the LARS score at 6, 9 and 12 months LARS difference score between inclusion and 6, 9 and 12-month follow-ups will be calculated using descriptive statistics and confidence intervals.
number of patients showing a change (reduction) of symptoms and consequences | 6, 9 and 12 months
  To assess the number of patients showing a change (reduction) of symptoms and consequences, as stated in the consensus definition at 6, 9 and 12 months The number and the proportion of patients with each item of the LARS international consensus definition at 6, 9 and 12 months will be calculated.
  Also, the proportion of patients who are considered as having no LARS at 6, 9 and 12 months will be calculated with a confidence interval.
Preference of the patient and reason for it | 12 month follow-up
  To assess the preference of the patient and reason for it Proportion of patients who stay on TAI treatment for TAI arm and proportion of patients from SOC arm whose tries and stay on TAI will be calculated using confidence intervals. Description of reasons will be also presented.
QoL with the EORTC QLQ-C30 and EORTC QLQ-CR29 at 12 month | 12-month follow-up
  to assess the QoL with the EORTC QLQ-C30 and EORTC QLQ-CR29 EORTC-QLQ-C30 and EORTC-QLQ-CR29 differences scores between inclusion and 12-month follow-ups will be calculated for each randomised arm using descriptive statistics and confidence intervals.
incontinence anal score at 12 months | 12-month follow-up
  Wexner difference score between inclusion and 12-month follow-up will be calculated for each randomised arm using descriptive statistics and confidence intervals.
  Also, statistical tests of superiority will be performed comparing Wexner differences between inclusion and 12-month follow-up between interventional arm and control arm
patient health organization and resources needed at 6, 9 and 12 months | 6, 9 and 12 months
  Data about quantity of organization and resources needed (professional activities, treatment, medical and specialize consultation, home helpers) will be presented using descriptive statistics

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Amiens-Picardie, Amiens
  - CHU Besançon, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - CHU Grenoble, La Tronche
  - CHU Timone, Marseille
  - CHU de NANTES, Hôtel Dieu, Nantes
  - CHU Bordeaux, GH Sud, Hôpital HAUT-LEVEQUE, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CHU Charles Nicolle - Rouen, Rouen